CLINICAL TRIAL: NCT05714163
Title: Effects of Ai Chi on Scapular Muscle Activation in Overhead Athletes With Scapular Dyskinesis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202208053RINA
Record Dates: First submitted 2022-10-12; First posted 2023-02-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Scapular Dyskinesis; Athletic Injuries; Muscle Weakness; Overuse Injury
Keywords: Ai Chi; Hydrotherapy; Scapular dyskinesis; Overhead athletes; muscle balance; kinetic chain
MeSH Terms: conditions — Athletic Injuries; Muscle Weakness; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scapular dyskinesis (SD) is common in overhead athletes and negatively influence the athletes' performance, increasing the risk of shoulder injury. The kinetic chain (KC) exercises for SD rehabilitation that emphasize importance of core strength and scapula stability during skillful performance. Ai Chi, the aquatic exercises performed in functional positions, which are adequate for power transfer of KC. This study will investigate the effect of KC-based water exercises, Ai Chi, on scapular muscles in overhead athletes with SD.

DETAILED DESCRIPTION:
The purpose of this study is to investigate muscle activations of the upper trapezius (UT), lower trapezius (LT), serratus anterior (SA), latissimus dorsi (LD), and muscle balance ratios of UT/LT, UT/SA I in overhead athletes with SD via KC-based exercise in water and on land. KC-based exercises including the movement patterns of Ai Chi which consist of shoulder flexion/ extension, horizontal abduction/ adduction, internal and external rotation, scapular protraction/retraction combined with spinal rotation.

ELIGIBILITY:
Inclusion Criteria:

* The participants are overhead athletes with scapular dyskinesis (SD) who played overhead sports activities at least 3 hours/week.

Exclusion Criteria:

* the individuals who have shoulder/neck pain in recent 3 months (VAS >7/10)
* severe shoulder trauma (the collision shoulder, shoulder sprains or strains)
* severe scoliosis (Cobb angle > 25 degrees)
* surgery of upper extremity (the shoulder, cervical spine and elbow) or cervical spine
* peripheral nerve injury or neurological disease (impaired sensation or motor function: numbness, tingle, muscle weakness)
* body mass index (BMI) >25
* infectious disease (upper respiratory tract infection, skin infection, etc.)

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are overhead athletes with scapular dyskinesis (SD) who played overhead sports activities at least 3 hours/week.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of maximal voluntary isometric contraction of upper trapezius (UT), lower trapezius (LT), serratus anterior (SA), latissimus dorsi (LD) | Through study completion, an average of 10 months
  The muscle activity of UT, LT, SA and LD of the dominant hand will be recorded for 3 trials of each exercises with 3-seconds concentric phase and 3-seconds eccentric phase. There is a 3-second rest between trails and one-minute rest between exercises.

SECONDARY OUTCOMES:
Muscle balance ratio of UT/SA | Through study completion, an average of 10 months
  The muscle balance ratio will be calculated to represent the conditions of these force couples in scapular region.
Muscle balance ratio of UT/LT | Through study completion, an average of 10 months
  The muscle balance ratio will be calculated to represent the conditions of these force couples in scapular region.

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-Jenq Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided